CLINICAL TRIAL: NCT00116428
Title: NAVISTAR® THERMOCOOL® Catheter for the Radiofrequency Ablation of Symptomatic Paroxysmal Atrial Fibrillation
Acronym: Afib IDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWI03130
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Heart Diseases; Arrhythmia; Atrial Fibrillation
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAVISTAR® THERMOCOOL® Catheter (Experimental)
  Interventions: Device: NAVISTAR® THERMOCOOL® Catheter
- Antiarrhythmic drug (Active Comparator)
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Device: NAVISTAR® THERMOCOOL® Catheter — The Biosense Webster NAVISTAR® THERMOCOOL® Diagnostic/Ablation Deflectable Tip Catheter is a luminal catheter with a deflectable tip designed to facilitate electrophysiological mapping of the heart and to transmit radiofrequency current to the catheter tip electrode for ablation purposes.
  Arms: NAVISTAR® THERMOCOOL® Catheter
Drug: Antiarrhythmic drug — Subjects randomized to the antiarrhythmic drug (control) arm will be prescribed to a not previously administered class I or class III antiarrhythmic drug that is currently approved in the U.S. for treating atrial fibrillation.
  Arms: Antiarrhythmic drug

SUMMARY:
This trial compares the safety and effectiveness of catheter ablation for PAF with antiarrhythmic drug therapy. The investigational catheter being studied is the NAVISTAR® THERMOCOOL® irrigated-tip catheter. At the time of this study, the NAVISTAR® THERMOCOOL® catheter was FDA-approved for commercial distribution in the U.S. for treating patients with Type I atrial flutter and drug refractory monomorphic ventricular tachycardia post myocardial infarction. The catheter was approved for use in Europe for endocardial ablation for treating cardiac arrhythmias.

ELIGIBILITY:
You may be eligible to participate in this study if you: Have failed to respond to drug treatment for your AFib, or find the side effects of your medication intolerable.

Inclusion Criteria

* Patients with symptomatic PAF who have had three (3) AF episodes in the six (6) months prior to randomization, one of which must be documented. Documentation may include electrocardiogram (ECG), transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip.
* Failure of at least one AAD for PAF [class I or III or AV nodal blocking agents such as beta blockers (BB) and calcium channel blockers (CCB)] as evidenced by recurrent symptomatic PAF, or intolerable side effects due to AAD.
* Signed Patient Informed Consent Form.
* Age 18 years or older.
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* Previous ablation for atrial fibrillation.
* Patients on amiodarone therapy at any time during the previous six (6) months.
* AF episodes that last longer than 30 days and are terminated via cardioversion.
* Any valvular cardiac surgical procedure.
* CABG procedure within the last 180 days (six months).
* Awaiting cardiac transplantation or other cardiac surgery within the next 360 days (12 months).
* Documented left atrial thrombus on imaging (e.g. TEE).
* History of a documented thromboembolic event within the past one (1) year.
* Diagnosed atrial myxoma.
* Presence of implanted ICD.
* Significant pulmonary disease, (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable).
* Acute illness or active systemic infection or sepsis.
* Unstable angina.
* Myocardial infarction within the previous 60 days (two months).
* LVEF < 40%.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation (i.e. heparin or warfarin).
* Contraindication to CT/MRA procedure.
* Life expectancy less than 360 days (12 months).
* Enrollment in an investigational study evaluating another device or drug.
* Uncontrolled heart failure or NYHA class III or IV heart failure.
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
* Presence of a condition that precludes vascular access.
* Left atrial size ≥ 50 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2007-10-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilber, MD, Principal Investigator — Loyola University
Locations (17):
- United States (13):
  - Marin General Hospital, Greenbrae, California
  - Florida Hospital, Orlando, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - St. Lukes Roosevelt Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Heart Hospital Baylor Plano Baylor Research Institute, Plano, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- Hospital Sao Paulo, São Paulo, Brazil
- Montreal Heart Institute, Montreal, Quebec, Canada
- Na Homolce Hospital, Prague, Motol, Czechia
- Hospital San Raffaele, Milan, Italy

REFERENCES:
- [Result] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Derived] Reynolds MR, Walczak J, White SA, Cohen DJ, Wilber DJ. Improvements in symptoms and quality of life in patients with paroxysmal atrial fibrillation treated with radiofrequency catheter ablation versus antiarrhythmic drugs. Circ Cardiovasc Qual Outcomes. 2010 Nov;3(6):615-23. doi: 10.1161/CIRCOUTCOMES.110.957563. Epub 2010 Oct 12. PMID 20940250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pivotal study was closed to enrollment on October 12, 2007 with a total of 167 subjects enrolled at 19 investigational sites (15 US and 4 outside US).
Groups:
- NAVISTAR® THERMOCOOL® Catheter: Subjects who were randomized to the THERMOCOOL group, i.e., to receive NAVISTAR® THERMOCOOL® Catheter at randomization. The Biosense Webster NAVISTAR® THERMOCOOL® Diagnostic/Ablation Deflectable Tip Catheter is a luminal catheter with a deflectable tip designed to facilitate electrophysiological mapping of the heart and to transmit radiofrequency current to the catheter tip electrode for ablation purposes.
- Antiarrhythmic Drug: The antiarrhythmic drug (control group) is defined as class I, class III or atrioventricular nodal blocking agents such as beta blocking agents (BB) or calcium channel blockers (CCB). During the two-week dosing period, the subject's medication was titrated up for maximum efficacy for the treatment of paroxysmal atrial fibrillation. The subject was maintained on the same drug for the rest of study time frame OR underwent a study ablation procedure after failing the effectiveness endpoint.
Period: Overall Study
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug
Started | 106 | 61
Underwent Study Ablation Procedure | 103 | 36
Completed | 103 | 56
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Did not meet inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug | Total
Number analyzed (Participants) | 106 | 61 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.3) | 56.1 (12.8) | 55.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 23 | 56
  Male | 73 | 38 | 111
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic | 1 | 0 | 1
    Native American | 1 | 0 | 1
    White | 103 | 61 | 164
    Arab ethnicity | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 7 | 5 | 12
  Canada | 5 | 3 | 8
  Czech Republic | 17 | 10 | 27
  Italy | 31 | 19 | 50
  United States | 46 | 24 | 70
Number of documented symptomatic Atrial Fibrillation episodes [Mean (Standard Deviation); unit: Number of episodes] — Number of symptomatic Atrial Fibrillation episodes during the last six months prior to study enrollment.
  Number of episodes | 62.3 (89.2) | 64.9 (98.0) | 63.24 (93.0)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Chronic Success of the NAVISTAR THERMOCOOL Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation (PAF)
Description: Chronic success was defined as freedom of documented symptomatic Atrial Fibrillation episodes based on electrocardiographic data and no changes in antiarrhythmic drugs (AAD) regimen during comparable evaluation periods for the THERMOCOOL and AAD (Control) groups through 12 and 9 months of follow-up, respectively.
Time Frame: The evaluation time frame for the THERMOCOOL catheter subjects is 91-361 days (12 months) post procedure; for Antiarrhythmic Drug Therapy subjects the time frame is 15-285 days (9 months) post procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug
Number analyzed (Participants) | 106 | 61
Percentage of participants | 66 | 16
Statistical Analysis 1: Comparison: NAVISTAR® THERMOCOOL® Catheter vs Antiarrhythmic Drug; The study null hypothesis is that the chronic success rates for the THERMOCOOL and AAD groups are equal; Test type: Superiority or Other; p < 0.001, Log Rank

2. Primary Outcome: The Percentage of Subjects Who Experienced Incidences of Early Onset (Within 7 Days of Ablation Procedure) Serious Catheter-related Adverse Events
Description: Catheter-related adverse events include death, myocardial infarction, pulmonary vein stenosis,diaphragmatic paralysis, atrio-esophageal fistula,transient ischemic attack,stroke,cerebrovascular accident, thromboembolism, pericarditis, cardiac tamponade,pericardial effusion,pneumothorax,atrial perforation,vascular access complications,pulmonary edema,hospitalization (initial and prolonged), and heart block.
Time Frame: Within 7 Days of Ablation Procedure
Population: Analysis population includes those enrolled subjects undergoing a study ablation procedure. A total of 139 underwent the procedure, including 36 AAD (control) group subjects who underwent the procedure after failing the effectiveness endpoint. The remaining 25 AAD (control) subjects didn't have the ablation procedure.
Measure: Number; unit: Percentage of Participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug
Number analyzed (Participants) | 139 | 25
Percentage of Participants | 10.1 | 0.0

3. Secondary Outcome: The Percentage of Subjects Who Achieved Acute Success.
Description: Acute success was defined as confirmation of entrance block in all targeted pulmonary veins. The study protocol considered subjects that had more than 2 AF ablation procedures within the 90 day blanking period immediately following their index study procedure or subjects that had additional ablation procedures greater than 80 days following their original study ablation procedure as acute failures.
Time Frame: 90 days post study procedure
Population: This analysis population is based on the first study ablation procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug
Number analyzed (Participants) | 103 | 36
Percentage of participants | 100 | 94

4. Secondary Outcome: Percentage of Subjects Who Experienced Atrial Fibrillation Recurrence During the Two-year Follow up.
Description: At the 2 year follow-up visit, Atrial Fibrillation recurrence was assessed by subject interview without documentation.
Time Frame: During the two years of post procedure
Population: Subjects who completed two years follow up
Measure: Number; unit: Percentage of Participants
Groups:
- Antiarrhythmic Drug Subjects Undergoing Ablation: Control Group Subjects underwent a study ablation procedure after failing the effectiveness endpoint.
- Antiarrhythmic Drug: The antiarrhythmic drug (control group) is defined as class I, class III or atrioventricular nodal blocking agents such as beta blocking agents (BB) or calcium channel blockers (CCB). During the two-week dosing period, the subject's medication was titrated up for maximum efficacy for the treatment of paroxysmal atrial fibrillation. The subject was maintained on the same drug for the rest of study time frame.
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug Subjects Undergoing Ablation | Antiarrhythmic Drug
Number analyzed (Participants) | 92 | 35 | 15
Percentage of Participants | 29.3 | 28.6 | 53.3

5. Secondary Outcome: Percentage of Subjects Responded to Each of the Four Health Status Categories.
Description: At the 2 year follow-up visit, Atrial Fibrillation recurrence was assessed by subject interview without documentation.
Time Frame: During the two years of post procedure
Population: Subjects who completed the two-year health survey.
Measure: Number; unit: Percentage of Participants
Groups:
- Antiarrhythmic Drug Subjects Undergoing Ablation: Control subjects underwent a study ablation procedure after failing the effectiveness endpoint.
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug Subjects Undergoing Ablation | Antiarrhythmic Drug
Number analyzed (Participants) | 92 | 35 | 15
Percentage of Participants
  Two-Year Health Status: Improved | 65.2 | 60.0 | 53.3
  Two-Year Health Status: Unchanged | 29.3 | 37.1 | 33.3
  Two-Year Health Status: Worsened | 5.4 | 2.9 | 6.7
  Two-Year Health Status: Missing | 0.0 | 0.0 | 6.7

ADVERSE EVENTS:
Groups:
- NAVISTAR® THERMOCOOL® Catheter: Subjects who were randomized to the THERMOCOOL group, i.e., to receive NAVISTAR® THERMOCOOL® Catheter at randomization; OR received the Catheter after failing the effectiveness endpoint. The Biosense Webster NAVISTAR® THERMOCOOL® Diagnostic/Ablation Deflectable Tip Catheter is a luminal catheter with a deflectable tip designed to facilitate electrophysiological mapping of the heart and to transmit radiofrequency current to the catheter tip electrode for ablation purposes.
- Antiarrhythmic Drug: The antiarrhythmic drug (control group) is defined as class I, class III or atrioventricular nodal blocking agents such as beta blocking agents (BB) or calcium channel blockers (CCB). During the two-week dosing period, the subject's medication was titrated up for maximum efficacy for the treatment of paroxysmal atrial fibrillation. The subject was maintained on the same drug for the rest of study time frame AND didn't undergo a study ablation procedure.
Arm/Group | NAVISTAR® THERMOCOOL® Catheter | Antiarrhythmic Drug
Serious Adverse Events (participants affected / at risk) | 25/139 | 0/25
Other Adverse Events (participants affected / at risk) | 23/139 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVISTAR® THERMOCOOL® Catheter (N=139) | Antiarrhythmic Drug (N=25)
Death (General disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Complication (Vascular disorders) | 5 (5) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization (Investigations) | 7 (7) | 0 (0)
Tearing of atrial septum (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemoptysis/Right Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Neoplasm/Kidney Nodule (Renal and urinary disorders) | 2 (2) | 0 (0)
Emergency Department Visit (Cardiac disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVISTAR® THERMOCOOL® Catheter (N=139) | Antiarrhythmic Drug (N=25)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Back pain (General disorders) | 3 (3) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Nausea, Vomiting/Rigors (Gastrointestinal disorders) | 2 (6) | 0 (0)
Neurologic Side Effects (Nervous system disorders) | 3 (3) | 0 (0)
Pericardial Effusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hematoma/Bleeding/groin pain (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is allowed to publish but must submit draft publication(s) to Biosense Webster, Inc. at least 30 days prior to submission for publication or presentation.